CLINICAL TRIAL: NCT03472144
Title: Gel-Sinuplasty for Chronic Rhinosinusitis With and Without Nasal Polyposis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: LifeBridge Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2397
Record Dates: First submitted 2017-12-15; First posted 2018-03-21 (Actual); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Chronic Sinusitis, Ethmoidal; Chronic Sinusitis - Ethmoidal Anterior; Chronic Sinusitis; Chronic Sinusitis - Ethmoidal, Posterior; Chronic Sinusitis, Sphenoidal; Chronic Sinusitis - Frontoethmoidal; Nasal Polyps; Nasal Polyp - Posterior
MeSH Terms: conditions — Nasal Polyps | interventions — Steroids; Anti-Bacterial Agents; Levofloxacin

STUDY DESIGN:
Intervention Model Description: This is a single-blinded Randomized Control Trial study, in which every patient receives active gel on one side and placebo on the other (L or R to be randomly selected).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Principle investigator will be non blinded and all others will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (12):
- CRSwNP - Subgrp 1(Momentasone - Right) (Experimental): Patients undergoing balloon sinuplasty will receive a gel loaded with steroids (Momentasone) only on right side and placebo on left side
  Interventions: Drug: gel loaded with steroids (momentasone)
- CRSwNP-Subgrp 2(Levofloxacin - Right) (Experimental): Patients undergoing balloon sinuplasty with receive a gel loaded with antibiotic (Levofloxacin) only on right side and placebo on left side
  Interventions: Drug: gel loaded with antibiotic (Levofloxacin)
- CRSwNP-Subgrp 3(Steroid/Antibotic Right) (Experimental): Patients undergoing balloon sinuplasty will receive a gel loaded with both steroids and antibiotic on right side and placebo on left side
  Interventions: Drug: gel loaded with both steroids and antibiotic
- CRSsNP - Subgrp 1 (Momentasone Right) (Experimental): Patients undergoing ballon sinuplasty will receive a gel loaded with steroids (Momentasone) only on right side and placebo on left side
  Interventions: Drug: gel loaded with steroids (momentasone)
- CRSsNP - Subgrp 2 (Levofloxacin Right) (Experimental): Patients undergoing balloon sinuplasty will receive a gel loaded with antibiotic (Levofloxacin) only on right side and placebo on left side
  Interventions: Drug: gel loaded with antibiotic (Levofloxacin)
- CRSsNP-Subgrp 3(Steroid/Antibiotic Right (Experimental): Patients undergoing balloon sinuplasty will receive a gel loaded with both steroids and antibiotic on right side and placebo on left side
  Interventions: Drug: gel loaded with both steroids and antibiotic
- CRSwNP - Subgrp 1 (Momentasone Left) (Active Comparator): Patients undergoing balloon sinuplasty will receive a gel loaded with steroids (Momentasone) only on left side and placebo on right side
  Interventions: Drug: gel loaded with steroids (momentasone)
- CRSwNP - Subgrp 2 (Levofloxacin Left) (Active Comparator): Patients undergoing balloon sinuplasty will receive a gel loaded with antibiotic (Levofloxacin) only left side and placebo on right side
  Interventions: Drug: gel loaded with antibiotic (Levofloxacin)
- CRSwNP-Subgrp 3(Steroid/Antibiotic Left) (Active Comparator): Patients undergoing balloon sinuplasty will receive a gel loaded with both steroids and antibiotic on left side and placebo on right side
  Interventions: Drug: gel loaded with both steroids and antibiotic
- CRSsNP - Subgrp 1 (Momentasone Left) (Active Comparator): Patients undergoing balloon sinuplasty will receive a gel loaded with steroids (Momentasone) only left side and placebo on right side
  Interventions: Drug: gel loaded with steroids (momentasone)
- CRSsNP - Subgrp 2 (Levofloxacin Left) (Active Comparator): Patients undergoing balloon sinuplasty will receive a gel loaded with antibiotic (Levofloxacin) only left side and placebo on right side
  Interventions: Drug: gel loaded with antibiotic (Levofloxacin)
- CRSsNP-Subgrp 3(Steroid/Antibiotic Left) (Active Comparator): Patients undergoing balloon sinuplasty will receive a gel loaded with both steroids and antibiotic on left side and placebo on right side
  Interventions: Drug: gel loaded with both steroids and antibiotic

INTERVENTIONS:
Drug: gel loaded with steroids (momentasone) — One of the purpose of this study is to evaluate the efficacy of a gel that actively releases local corticosteroids (momentasone) after balloon sinuplasty for chronic sinusitis patients.
  Other Names: Momentasone
  Arms: CRSsNP - Subgrp 1 (Momentasone Left); CRSsNP - Subgrp 1 (Momentasone Right); CRSwNP - Subgrp 1 (Momentasone Left); CRSwNP - Subgrp 1(Momentasone - Right)
Drug: gel loaded with antibiotic (Levofloxacin) — One of the purpose of this study is to evaluate the efficacy of a gel that actively releases local antibiotic(levofloxacin) after balloon sinuplasty for chronic sinusitis patients.
  Other Names: Levofloxacin
  Arms: CRSsNP - Subgrp 2 (Levofloxacin Left); CRSsNP - Subgrp 2 (Levofloxacin Right); CRSwNP - Subgrp 2 (Levofloxacin Left); CRSwNP-Subgrp 2(Levofloxacin - Right)
Drug: gel loaded with both steroids and antibiotic — One of the purpose of this study is to evaluate the efficacy of a gel that actively releases local both steroids (momentasone)and antibiotic(levofloxacin) after balloon sinuplasty for chronic sinusitis patients.
  Other Names: Momentasone, Levofloxacin
  Arms: CRSsNP-Subgrp 3(Steroid/Antibiotic Left); CRSsNP-Subgrp 3(Steroid/Antibiotic Right; CRSwNP-Subgrp 3(Steroid/Antibiotic Left); CRSwNP-Subgrp 3(Steroid/Antibotic Right)

SUMMARY:
To assess the efficacy of intra-sinus installation of a poloxamer gel that releases antibiotics and corticosteroids topically after balloon sinuplasty in chronic sinusitis patients with or without polyps. This is a single-blinded Randomized Control Trial study, in which every patient receives active gel on one side and placebo on the other (L or R to be randomly selected).

DETAILED DESCRIPTION:
STUDY DESIGN This is a single-blinded Randomized Control Trial study, in which every patient receives active gel on one side and placebo on the other (L or R to be randomly selected). Sixty patients will be included in this study. These are patients undergoing balloon sinuplasty for Chronic sinusitis with and without polyps.

As the patients will enter the study- they will be divided into Chronic sinusitis with Polyps (CRSwNP) and Chronic rhinosinusitis without polyps (CRSsNP). Each patient will be assigned in chronological order as they will join the study.

For each group, all even numbered patients will receive the active gel application on right side and all odd number patients will receive the active gel on left side.

Then patient selection for CRSwNP and CRSsNP will be as such Each group will have 3 subgroups. Subgroup 1- gel will be loaded with steroids only Subgroup 2- gel will be loaded with antibiotic (Levaquin) only Subgroup 3- gel will be loaded with both steroids and antibiotic CRSwNP group with right side gel application Subgroup 1- patient number- 1,7,13,19,25 Subgroup 2- patient number- 3,9,15,21,27 Subgroup 3- patient number- 5,11,17,23,29 CRSwNP group with left side gel application Subgroup 1- patient number- 2,8,14,20,26 Subgroup 2- patient number- 4,10,16,22,28 Subgroup 3- patient number- 6,12,18,24,30

A similar patient randomization will be done with the CRSsNP group

Surgery will consist of plain balloon sinuplasty or hybrid balloon sinuplasty with removal of ethmoids polypss using a Blakesley forceps. During surgery, and immediately after removal of diseased mucosa, 5 ccs of an active poloxamer gel containing the antibiotic or corticosteroids or both will be instilled inside the ethmoid/ maxillary sinus/frontal cavities on one side using either the balloon catheter or as a curved suction tip. The same procedure is performed in the other side, this time with instillation of plain gel without antibiotic or corticosteroids (placebo).

The purpose of the study is to assess the efficacy of intra-sinus installation of a poloxamer gel that releases antibiotics and corticosteroids topically after balloon sinuplasty in chronic sinusitis patients with or without polyps. The assessment of the healing process will be done at the end of one month then at two, three and six months. Total number of visits would be 8 including the operation day.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic sinusitis symptoms with or without polyps
2. Trial of at least 2 courses of oral antimicrobial treatment without significant improvement
3. CAT scan showing evidence of bilateral symmetric chronic sinusitis with or without polypss
4. Endoscopic confirmation of CRS

Exclusion Criteria:

1. Minor (Less than <18 years of age).
2. Pregnant and breastfeeding women.
3. Allergy to specific antibiotics
4. Patient currently taking oral corticosteroids.
5. Patient currently taking oral antibiotics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-07-07 (Actual); Primary Completion 2019-07-07 (Estimated); Study Completion 2019-12-07 (Estimated)

PRIMARY OUTCOMES:
Clinical improvement reported on SNOT-22 questionnaire | The total duration of the actual study is 30 months, and the follow up period per patient will 6 months postoperatively.
  Assessment of the healing process will be done at the end of one month then at two, three and six months. Total number of visits would be 8 including the operation day.
Improvement in the Lund-Kennedy endoscopic appearance scores. Improvement in the Lund-Kennedy endoscopic appearance scores | The total duration of the actual study is 30 months, and the follow up period per patient will 6 months postoperatively.
  Assessment of the healing process will be done at the end of one month then at two, three and six months. Total number of visits would be 8 including the operation day. Polyps (left, right) Edema (left, right) Discharge (left, right) Scarring (left, right) Crusting (left, right)
  Scoring:
  Polyps on left side - (0 absent, 1 polyps in middle meatus, 2 polyps beyond middle meatus) Polyps on right side - (0 absent, 1 polyps in middle meatus, 2 polyps beyond middle meatus) Edema, scarring and crusting on left side (0 absent, 1 mild, 2 severe) Edema, scarring and crusting on right side (0 absent, 1 mild, 2 severe) Discharge on left side (0, no discharge, 1 clear, thin discharge, 2 thick purulent discharge) Discharge on right side (0, no discharge, 1 clear, thin discharge, 2 thick purulent discharge)

SECONDARY OUTCOMES:
Radiological improvement of the Lund-Mackay score | The total duration of the actual study is 30 months, and the follow up period per patient will 6 months postoperatively.
  Assessment of the healing process will be done at the end of one month then at two, three and six months. Total number of visits would be 8 including the operation day. Paranasal sinuses Right Left Maxillary (0, 1, 2) Anterior Ethmoid (0, 1, 2) Posterior Ethmoid (0, 1, 2) Sphenoid (0, 1, 2) Frontal (0, 1, 2)
  * Ostiomeatal complex (0, 2) Total Note: 0- without abnormalities; 1- partial opacification; 2-total opacification
  * 0-no obstruction; 2-obstructed

CONTACTS AND LOCATIONS:
Overall Officials: Alan H. Shikani, MD, Principal Investigator — Sinai Hospital of Baltimore
Locations (1):
- Sinai Hospital of Baltimore, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
undecided so far

REFERENCES:
- [Background] Rosenfeld RM, Andes D, Bhattacharyya N, Cheung D, Eisenberg S, Ganiats TG, Gelzer A, Hamilos D, Haydon RC 3rd, Hudgins PA, Jones S, Krouse HJ, Lee LH, Mahoney MC, Marple BF, Mitchell CJ, Nathan R, Shiffman RN, Smith TL, Witsell DL. Clinical practice guideline: adult sinusitis. Otolaryngol Head Neck Surg. 2007 Sep;137(3 Suppl):S1-31. doi: 10.1016/j.otohns.2007.06.726. PMID 17761281
- [Background] Vaughan WC. Review of balloon sinuplasty. Curr Opin Otolaryngol Head Neck Surg. 2008 Feb;16(1):2-9. doi: 10.1097/MOO.0b013e3282f5e955. PMID 18197013
- [Background] Hopkins C, Browne JP, Slack R, Lund V, Brown P. The Lund-Mackay staging system for chronic rhinosinusitis: how is it used and what does it predict? Otolaryngol Head Neck Surg. 2007 Oct;137(4):555-61. doi: 10.1016/j.otohns.2007.02.004. PMID 17903570
- [Background] Alves DA, Machado D, Melo A, Pereira RF, Severino P, de Hollanda LM, Araujo DR, Lancellotti M. Preparation of Thermosensitive Gel for Controlled Release of Levofloxacin and Their Application in the Treatment of Multidrug-Resistant Bacteria. Biomed Res Int. 2016;2016:9702129. doi: 10.1155/2016/9702129. Epub 2016 Sep 5. PMID 27689094
- [Background] Li C, Gu J, Mao X, Ao H, Yang X. Preparation of levofloxacin thermo-sensitive gel and clinical application in the treatment of suppurative otitis media. Acta Otolaryngol. 2014 May;134(5):468-74. doi: 10.3109/00016489.2013.878473. Epub 2014 Mar 6. PMID 24597493
- [Background] Dumortier G, Grossiord JL, Agnely F, Chaumeil JC. A review of poloxamer 407 pharmaceutical and pharmacological characteristics. Pharm Res. 2006 Dec;23(12):2709-28. doi: 10.1007/s11095-006-9104-4. Epub 2006 Nov 11. PMID 17096184
- [Result] Shikani AH, Chahine KA, Alqudah MA. The rhinotopic protocol for chronic refractory rhinosinusitis: how we do it. Clin Otolaryngol. 2010 Aug;35(4):329-32. doi: 10.1111/j.1749-4486.2010.02157.x. No abstract available. PMID 20738346
- [Result] Shikani AH, Chahine KA, Alqudah MA. Rhinotopic therapy for refractory chronic rhinosinusitis: a study of 20 cases. Ear Nose Throat J. 2014 Apr-May;93(4-5):E48-54. PMID 24817242
- [Result] Shikani AH, Kourelis K, Rohayem Z, Basaraba RJ, Leid JG. Topical gel therapy for sinonasal polyposis in Samter's triad: preliminary report. Ann Otol Rhinol Laryngol. 2012 Nov;121(11):719-24. doi: 10.1177/000348941212101104. PMID 23193904